CLINICAL TRIAL: NCT07310043
Title: Creatine Intervention in Older Adults to Improve Perioperative Brain Health
Brief Title: Creatine and Perioperative Brain Health
Acronym: CREATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Susana Vacas, MD, PhD, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025P002111
Record Dates: First submitted 2025-12-12; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Neurocognitive Disorders; Postoperative Delirium
Keywords: Perioperative Brain Health; Creatine; Perioperative Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders; Emergence Delirium | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients under creatine monohydrate intervention (Experimental)
  Interventions: Dietary Supplement: Creatine monohydrate

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — Participants will receive creatine supplementation before surgery

SUMMARY:
The goal of this study is to understand the effects of oral creatine supplementation in the perioperative period. Creatine is commonly used to enhance athletic performance, but it can also have positive effects on the brain. Since surgery can lead to alterations in thinking, memory, and attention patterns in some patients, we will assess whether creatine can be protective against these changes in older adults undergoing surgery.

DETAILED DESCRIPTION:
Surgical interventions, while often necessary, are associated with substantial postoperative morbidity, particularly among older adults. Perioperative neurocognitive disorders (PND), characterized by changes in memory patterns in the perioperative period and are among the most common surgical complications in aging populations. Beyond their considerable economic burden, estimated to exceed $30 billion annually, PND impose profound immediate consequences for patients and caregivers and is associated with long-term adverse outcomes, including an increased risk of dementia. Despite their high prevalence and clinical impact, effective, scalable, and easily implementable preventive strategies for PND remain limited.

Creatine plays a critical role in supporting the brain's high metabolic demands, and its homeostasis may be disrupted during periods of physiological stress such as anesthesia and surgery. Creatine supplementation has demonstrated neuroprotective effects in other high-stress conditions. However, its potential to mitigate perioperative cognitive vulnerability has not been previously investigated. This study will evaluate creatine supplementation as a novel protective strategy to reduce the risk of PND in older adults undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* History of creatine deficiency disorders
* Severe neurologic or psychiatric diseases
* History of stroke or head trauma
* Obesity (BMI ≥ 30 kg.m-²), kidney or liver disease

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Preoperative cognitive function assessed with the Montreal Cognitive Assessment (MoCA) | Within three weeks before surgery
  The MoCA is a validated tool to assess cognitive function. Scores range from 0-30, with higher scores representing better cognitive function
Postoperative cognitive function assessed with the Montreal Cognitive Assessment (MoCA) | Within one month after surgery
  The MoCA is a validated tool to assess cognitive function. Scores range from 0-30, with higher scores representing better cognitive function
Postoperative cognitive function assessed with the Montreal Cognitive Assessment (MoCA) | Within three months after surgery
  The MoCA is a validated tool to assess cognitive function. Scores range from 0-30, with higher scores representing better cognitive function
Postoperative delirium assessed with the Confusion Assessment Method | Up to 7 days after surgery
  The CAM is a validated tool to detect postoperative delirium